CLINICAL TRIAL: NCT02261987
Title: Role of Resistive Inspiratory Manoeuvres During Bronchial Drainage Session in Cystic Fibrosis: a Randomized Crossover Trial
Brief Title: Resistive Inspiratory Manoeuvre as Airway Clearance Technique in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FR_FQ- 013
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis
Keywords: Autogenic drainage; Resistive inspiratory manoeuvre; Computerized respiratory sounds; Airway clearance techniques; Mucus clearances
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autogenic drainage (AD) (Active Comparator): Patients will perform the autogenic drainage technique following the Chevallier and Agostini recommendations.
  Interventions: Other: Autogenic drainage (AD)
- Resistive inspiratory manoeuvre (RIM) (Active Comparator): Patients will perform the repetitive inspiratory manoeuvers by breathing through a fixed resistance (Power Breathe device, model KH1) . Each session will comprise to cycles of 5 inspiratory breaths (60% of maximal inspiratory pressure). Patients will be stay in both lateral decubitus position (15 min per side).
  Interventions: Other: Resistive inspiratory manoeuvre (RIM)
- Resistive inspiratory manoeuvre+autogenic drainage (Active Comparator): First, patients will perform the resistive inspiratory manoeuvre during 10 minutes (5 min per side). Right after, patients will perform the autogenic drainage during 20 minutes.The instructions will be similar to described previously.
  Interventions: Other: Resistive inspiratory manoeuvre+autogenic drainage

INTERVENTIONS:
Other: Autogenic drainage (AD) — It will be apply in one only session. The time spent during this bronchial drainage session will be 30 minutes All patients will perform all interventions in a randomized order.
  Arms: Autogenic drainage (AD)
Other: Resistive inspiratory manoeuvre (RIM) — It will be apply in one only session. The time spent during this bronchial drainage session will be 30 minutes All patients will perform all interventions in a randomized order.
  Arms: Resistive inspiratory manoeuvre (RIM)
Other: Resistive inspiratory manoeuvre+autogenic drainage — It will be apply in one only session. The time spent during this bronchial drainage session will be 30 minutes All patients will perform all interventions in a randomized order.
  Arms: Resistive inspiratory manoeuvre+autogenic drainage

SUMMARY:
This trial aims to analyze whether the resistive inspiratory manoeuvre (RIM) performed previously to autogenic drainage (AD) technique improves the effectiveness in terms of mucus clearance during a typical bronchial drainage session in adults, stable CF patients.

DETAILED DESCRIPTION:
It is a multicenter study. 4 different Spain Cystic Fibrosis Foundations are included in the study (Madrid, Valencia, Murcia and Aragón). All patients will perform three different arms of treatment in a crossover randomization. Each arm of treatment will be apply only in one session. The wash-out period will be one week. Before starting the trial, all patients will perform a control session without any intervention, only the outcome measures will be assess.

During the study period the patients' pharmacological treatment remained unchanged

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis (CF) diagnosed ( established by genotype or sweat sodium>70 mmol/l or sweat chloride of>60 mmol/l)
* Clinically stable at time of study entry (defined as no requirement for antibiotics or change in respiratory medication in the preceding 4 wk);
* Chronic sputum production, at least ≥ 15 ml /24h
* Familiar and trained in the use of autogenic drainage technique (at least 6 months) and resistive inspiratory manoeuvre (at least three previous sessions)
* To be able to provide written, informed consent

Exclusion Criteria:

* Lung function: Forced expiratory volume in 1 second < 30 % pred . ; Forced vital capacity < 40 % pred.
* Active haemoptysis during the previous month
* Supplemental oxygen or non-invasive ventilation (NIV)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Wet sputum production | 24 hours
  24h wet sputum production (g) after bronchial drainage session

SECONDARY OUTCOMES:
Wet sputum production | 30 minutes
  Wet sputum production (g) during bronchial drainage session
Computerized respiratory sounds | 30 minutes
  Adventitous respiratory sounds: crackles and wheezes
Lung function (simply spirometry) | 30 minutes
  Forced expiratory volume at 1 second, Forced vital capacity, Forced expiratory flow 25-75
Patients´ perception | 30 minutes
  Visual analogical scale

OTHER OUTCOMES:
Pulse-oximetry, heart rate and dyspnea | 30 minutes
  Safety and tolerability of session

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Herrero, Msc, Principal Investigator — Universidad San Jorge
Locations (4):
- Spain (4):
  - Cystic Fibrosis Association, Madrid, Madrid
  - Cystic Fibrosis Association, Murcia, Murcia
  - Cystic Fibrosis Association, Valencia, Valencia
  - Universidad San Jorge, Zaragoza, Zaragoza

REFERENCES:
- [Result] Chatham K, Ionescu AA, Nixon LS, Shale DJ. A short-term comparison of two methods of sputum expectoration in cystic fibrosis. Eur Respir J. 2004 Mar;23(3):435-9. doi: 10.1183/09031936.04.00084904. PMID 15065835